CLINICAL TRIAL: NCT06617169
Title: Open Label, Phase 1a, Dose-Escalation Study Evaluating the Safety of Fractionated MNPR-101-PCTA-177Lu Dosing in the Treatment of Solid Tumor Cancers
Brief Title: Dose-Escalation of MNPR-101-PCTA-177Lu in Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Monopar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MNPR101-Lu-1-01
Record Dates: First submitted 2024-09-18; First posted 2024-09-27 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Solid Tumor, Adult; Bladder Cancer; Urothelial Carcinoma; Triple-negative Breast Cancer; Lung Cancer; Colorectal Cancer; Gastric Cancer; Ovarian Cancer; Pancreatic Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell; Triple Negative Breast Neoplasms; Lung Neoplasms; Colorectal Neoplasms; Stomach Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will be dosed in cohorts of two, starting at Dose Level 1. TITE-BOIN evaluates the number of participants that have been dosed at a given dose level and their outcomes and determines if the next cohort should stay at the same dose, increase dose, or decrease dose using a predetermined rule.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Level 0 - MNPR-101-PCTA-177Lu 480 MBq (Experimental)
  Interventions: Drug: MNPR-101-PCTA-177Lu
- Level 1 - MNPR-101-PCTA-177Lu 960 MBq (Experimental)
  Interventions: Drug: MNPR-101-PCTA-177Lu
- Level 2 - MNPR-101-PCTA-177Lu 1440 MBq (Experimental)
  Interventions: Drug: MNPR-101-PCTA-177Lu
- Level 3 - MNPR-101-PCTA-177Lu 1920 MBq (Experimental)
  Interventions: Drug: MNPR-101-PCTA-177Lu
- Level 4 - MNPR-101-PCTA-177Lu 2240 MBq (Experimental)
  Interventions: Drug: MNPR-101-PCTA-177Lu

INTERVENTIONS:
Drug: MNPR-101-PCTA-177Lu — MNPR-101-PCTA-177Lu administered intravenously over approximately 20 minutes, followed by a normal saline flush. Dosing will occur on Cycle 1 Day 1, Cycle 1 Day 15, and Cycle 2 Day 1.

SUMMARY:
This is an open-label, uncontrolled, multi-center, phase 1a MNPR-101-PCTA-177Lu dose-escalation study in patients with solid tumor cancers. Patients must have participated in the imaging study MNPR-101-D001 (actively recruiting, diagnostic study of MNPR-101-DFO*-89Zr).

* TITE-BOIN will be used to objectively determine dose increase, no dose change, or dose decrease for each group of two patients.
* The treatment period consists of two 12-week cycles. Patients will receive three equal fractions of MNPR-101-PCTA-177Lu with radioactivity ranging from 480-2240 MBq on each of Cycle 1 Day 1, Cycle 1 Day 15, and Cycle 2 Day 1 (12 weeks after Cycle 1 Day 1).
* Patients will be followed for 12 weeks after their last dose of MNPR-101-PCTA-177Lu.
* Patients will be imaged at specific timepoints during the study.

DETAILED DESCRIPTION:
This Phase 1a study will enroll qualified participants from the MNPR-101-D001 imaging study. Patients will receive three equal doses of MNPR-101-PCTA-177Lu, dose-escalating in cohorts of two starting at Dose Level 1 (960 MBq).On Cycle 1 Day 1, Cycle 1 Day 15, and Cycle 2 Day 1, patients will receive a 20-minute intravenous infusion of MNPR-101-PCTA-177Lu consisting of an antibody with radioactivity ranging from 480-2240 MBq (Dose Levels 0-4).

This study employs a Time-to-Event Bayesian Optimal Interval Design (TITE-BOIN). Dosing of subsequent cohorts will escalate, stay, or de-escalate based on TITE-BOIN predetermined, fixed dose escalation / de-escalation rules.

Any hematologic event must be ≤ Grade 1 for dosing to occur, i.e., patients with an active ≥ Grade 2 hematologic event may not be dosed. Any patient experiencing a ≥ Grade 2 allergic reaction during or immediately following infusion will not receive further treatment. Patients experiencing a DLT, at least possibly related to MNPR-101-PCTA-177Lu and occurring within 6 weeks of C1D1, will not receive any further doses. C1D15 and C2D1 doses may be delayed for up to 14 days for specified adverse events.

All subjects will undergo SPECT imaging on Cycle 1 Day 8 and Cycle 2 Day 8. CT scans will occur on Cycle 1 Day 43, Cycle 2 Day 1, and Cycle 2 Day 43; a baseline CT scan must be provided. These will allow for the assessment of tumor SUVs, as well as the radiologic response rate by RECIST 1.1.

Patients will be followed for safety for 12 weeks following the last dose of MNPR-101-PCTA-177Lu.

ELIGIBILITY:
Inclusion Criteria:

1. Participated in the MNPR-101-D001 study.
2. Females of childbearing potential must have a negative serum pregnancy test at time of screening and a negative urine pregnancy test on Day 1 prior to study drug administration if screening is >7 days prior to Day 1. A rapid serum pregnancy test result performed as standard of care will be accepted if available.
3. Both males and females must agree to use highly effective contraceptive precautions if conception is possible during the dosing period and up to 3 months after dosing.
4. Female patients who are lactating must agree to discontinue breastfeeding prior to the dose of study drug and must refrain from breastfeeding for 3 months following the last dose of study drug.

Exclusion Criteria:

1. Chemotherapy, radiotherapy (other than short cycle of palliative radiotherapy), or immunotherapy within 14 days prior to administration of MNPR-101-PCTA-177Lu.
2. Continuing ≥ Grade 3 adverse reactions from prior systemic therapy (Common Terminology Criteria for Adverse Events [CTCAE] version 5.0).
3. Prior treatment with any radiopharmaceutical or investigational agents within 4 weeks or 5 half-lives, whichever is longer, prior to administration of the first dose of MNPR-101-PCTA-177Lu other than MNPR-101-DFO*-89Zr.
4. Have evidence of impaired organ function at Screening and prior to dosing, particularly:

   • Bone marrow: i. Platelets ≤150×10^9/L. ii. Absolute neutrophil count ≤1.5×10^9/L. iii. Hemoglobin <9g/dL (no red blood cell transfusion in the previous 4 weeks).

   • Liver function: i. AST/ALT >3xULN (institutional upper limits of normal) OR >5×ULN for patients with liver metastases.

   ii. Bilirubin >1.5xULN OR >3xULN for patients with known Gilbert's Syndrome.

   • Renal function: i. eGFR ≤45 mL/min determined using BSA-adjusted Chronic Kidney Disease Epidemiology Collaboration CKD-EPI 2021 formula [https://www.kidney.org/professionals/kdoqi/gfr_calculator].
5. Safety event of significance in MNPR-101-D001 study:

   1. a related CTCAE Grade 4 hematologic or hepatologic event
   2. a related CTCAE Grade 3 hematologic or hepatologic event which lasted >30 days
6. Unacceptable value for projected organ dose based upon dosimetry from the MNPR-101-D001 study that exceeds safe absorbed dose limits, as determined by Monopar.
7. Other serious, non-malignant diseases (e.g., renal, hepatic, or hematologic) that may interfere with objectives of the study, safety, or compliance, as judged by the investigator.
8. Cognitive impairment or contraindications that may compromise ability to give informed consent or comply with requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Identify the dose-limiting toxicities (DLTs) of fractionated MNPR-101-PCTA-177Lu dosing and their frequency | For 6 weeks after the first dose
  Dose-limiting toxicities (DLT) are at least possibly related to MNPR-101-PCTA-177Lu and occur within 6 weeks of C1D1. Participants experiencing a DLT will not receive any further doses. Participants will continue study participation through the 12-week post final dose Safety Visit.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] of fractionated MNPR-101-PCTA-177Lu dosing | From dosing to the End of Study at 24 weeks
  The safety profile of MNPR-101-PCTA-177Lu will be determined through assessment of adverse event (AE) type, incidence, severity, time of appearance, and related causes (detected by physical explorations and laboratory tests). Adverse events will be graded and tabulated using NCI CTCAE v5.0.

SECONDARY OUTCOMES:
Assessment radiologic response rate by RECIST 1.1 | Every 6 weeks after initial dose
  Radiologic response rate will be determined by RECIST 1.1 via CT scans every 6 weeks (3 timepoints).
Assessment of radiologic response rate by PERCIST 1.0 | At 12 weeks after first dose (End of Cycle 1) and at 12 weeks after final dose (Safety Visit)
  Radiologic response rate determined by PERCIST 1.0 via PET scans (non-CT measurable participants)
Assess Radioactivity in whole blood and plasma following each fractionated MNPR-101-PCTA-177Lu dose | for 2 weeks after each dose
  Radioactivity in whole blood and plasma for each fractionated MNPR-101-PCTA-177Lu are projected via time-corrected gamma counts.
To determine the maximum administered dose (MAD) for fractionated MNPR-101-PCTA-177Lu dosing | 6 weeks after the first dose
  The maximum administered dose will be determined by the highest dose of MNPR-101-PCTA-177Lu not eliminated by TITE-BOIN.

CONTACTS AND LOCATIONS:
Locations (1):
- Melbourne Theranostic Innovation Centre (MTIC), North Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No